CLINICAL TRIAL: NCT02641470
Title: Clinical Trial to Investigate the Effect of DA9301 on Tablet Computer-induced Asthenopia in Humans
Brief Title: The Effect of DA9301 on Tablet Computer-Induced Asthenopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namyi Gu (Other)
Responsible Party: Sponsor-Investigator, Namyi Gu, Assistant professor, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA9301_01
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Asthenopia
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA9301 (Experimental): Orally administration of DA9301 (Vaccinium uliginosum extract) pills (1000 mg/day) for 4 weeks.
  Interventions: Dietary Supplement: DA9301 (Vaccinium uliginosum extract)
- Placebo (Placebo Comparator): Orally administration of placebo pills (1000 mg/day) for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DA9301 (Vaccinium uliginosum extract)
  Arms: DA9301
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Asthenopia or eye strain describes nonspecific symptoms of an eye when it is tired from intensive work. Vaccinium uliginosum is a flowering plant in the genus Vaccinium. This plant is native to cool temperature regions of the Northern Hemisphere. Considering its antioxidative ingredients, the extract of Vaccinium uliginosum is expected to play a significant role in treating various ocular pathologies. The investigators performed a randomized, case-controlled study in healthy subjects and investigated the protective effect of Vaccinium uliginosum extract (DA-9301) on tablet computer-induced asthenopia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject aged 20 to 65 years with more than 2 hours of daily use of a smart phone or computer including a tablet and television

Exclusion Criteria:

1. Ocular disease in either eye

   * Ocular surface disease
   * Best corrected visual acuity < 20/30
   * Intraocular pressure > 21 mmHg
   * Optical coherence tomography proven retinal nerve fiber defect
   * Significant cataract (lens opacities classification system III)
   * Significant entropion or ectropion
   * Significant tear drainage problem proved with fluorescein dye dilution test
2. Soft or Hard contact lens use 3 or more days a week
3. History of oral intake of health supplement designed to improve asthenopia within 4 weeks before participating this study
4. Pregnant woman
5. Systemic disease

   * Uncontrolled hypertension (systolic /diastolic blood pressure > 140/90mmHg)
   * Uncontrolled diabetes mellitus (fasting blood glucose level > 180mg/dL)
   * Rheumatoid arthritis
   * Malignant disease
   * Active hepatitis (type B and C)
   * Acute or chronic infectious disease
   * Renal disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change of the modified questionnaire scores proposed by Ames et al. | before and immediately after tablet computer use on Day 0 and Day 29 (deviation window: Day 21-31)

CONTACTS AND LOCATIONS:
Overall Officials: Choul Yong Park, MD, PhD, Principal Investigator — oph0112@gmail.com

REFERENCES:
- [Derived] Park CY, Gu N, Lim CY, Oh JH, Chang M, Kim M, Rhee MY. The effect of Vaccinium uliginosum extract on tablet computer-induced asthenopia: randomized placebo-controlled study. BMC Complement Altern Med. 2016 Aug 18;16:296. doi: 10.1186/s12906-016-1283-x. PMID 27538497